CLINICAL TRIAL: NCT02393092
Title: A Youth Violence Prevention Initiative: A VCUHS and Boys and Girls Club of Metro Richmond Initiative
Brief Title: Violence Prevention Study for Youth Age 10-15
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was determined that internal resources to support this population would be better utilized in other Injury and Violence Prevention Programs.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Boys and Girls Clubs of Metro Richmond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20002499
Record Dates: First submitted 2015-03-03; First posted 2015-03-19 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Violence, Non-accidental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BVA Only (Experimental): Study participants in this arm will only receive a Brief Violence Awareness (BVA) intervention.
  Interventions: Behavioral: Brief Violence Awareness
- BVP Only (Experimental): Study participants in this arm will only receive a Brief Violence Prevention (BVP) intervention.
  Interventions: Behavioral: Brief Violence Prevention
- Emerging Leaders plus BVP (Experimental): Study participants in this arm will participate in the Emerging Leaders: East End curriculum at the Boys and Girls Club of Metro Richmond, Martin Luther King Jr. Middle School site. They will also receive a Brief Violence Prevention (BVP) intervention.
  Interventions: Behavioral: Brief Violence Prevention; Behavioral: Emerging Leaders: East End curriculum

INTERVENTIONS:
Behavioral: Brief Violence Awareness — The Brief Violence Awareness (BVA) will consist of a packet of information about violence prevention and local community resources.
  Arms: BVA Only
Behavioral: Brief Violence Prevention — The Brief Violence Prevention (BVP) will be a psycho-educational intervention administered by a case manager that will include an interactive discussion with youth regarding resources for remaining safe and preventing violence. The intervention will address the concerns and questions of youth and youth will be given information on how to access community based resources if needed.
  Arms: BVP Only; Emerging Leaders plus BVP
Behavioral: Emerging Leaders: East End curriculum — The Emerging Leaders: East End curriculum focuses on positive youth development and education, which includes an emphasis on health careers. The curriculum will be administered at the Boys and Girls Club of Metro Richmond, Martin Luther King Middle School site.
  Arms: Emerging Leaders plus BVP

SUMMARY:
This study will evaluate the effectiveness of a hospital-community based violence prevention pilot study designed to increase protective factors and reduce negative risk factors associated with violence of children aged 10-15. Behaviors and attitudes that relate to violence and behavior change will be assessed through a series of questionnaires administered in an interview format. Assessments will occur every nine weeks. Additionally, objective long term measures for violence related hospital visits, delinquency, and educational development will be obtained.

The study will include the following interventions:

1. Brief violence prevention (BVP): a case manager administered psycho-educational intervention that will include an interactive discussion with youth regarding resources for remaining safe and preventing violence. The intervention will address the concerns and questions of youth and youth will be given information on how to access community based resources if needed.
2. Brief violence awareness (BVA): a packet of information about violence prevention and local community resources.
3. Emerging Leaders: East End: a semester (17 weeks) long curriculum based positive youth development education program held at the Boys and Girls Club of Metro Richmond, Martin Luther King Middle School site that includes case management to ensure continued engagement and participation.

Specifically, it is hypothesized that:

1. Participants will report more positive youth behaviors as compared to their initial assessment.
2. Participants will report lower levels of risky youth behaviors compared to their initial assessment.
3. Participants will report increased interest in and knowledge of health professions.
4. Participants will report reduced levels of delinquency compared to their initial assessment.
5. Participants will report a reduction in the number of violence related hospital visits compared to the general 23223 population.
6. Hospital data will show a reduction in violence related activities that led to hospital visits, or delinquent behavioral involvement.

DETAILED DESCRIPTION:
The study will include children living in the 23223 zip code of the City of Richmond, who attend Martin Luther King Middle School, and who are between the ages 10-15. The study will recruit from two sites. These sites include the Pediatric Emergency Department at VCU Medical Center and the Boys and Girls Club of Metro Richmond, Martin Luther King Middle School site. Upon recruitment, consent, and assessment, the children will receive either 1) a BVP only, 2) a BVA only or 3) a BVP as well as participation in a semester-long positive youth development program called Emerging Leaders: East End. The randomization process among all three groups will be done through sequential selection. Youth will be assigned to one of the three groups on a rotating, sequential basis as they enroll.

The study will assess behaviors, attitudes, family function, violence exposure, mental health, medical needs and service needs. The study will compare within group differences between a group that receives the BVP intervention and attends the Emerging Leaders: East End program, one that only receives the BVP intervention, one that receives a BVA intervention package only and one that receives the BVA or BVP and attends the Boys and Girls club but does not participate in the Emerging Leaders: East End program.

All groups will take an assessment every nine weeks through Grade 12 or until youth end their participation in this study. The assessment tool includes topics such as exposure to violence, family functioning and mental health. Case managers will administer the assessment.

Within the overall goal of reducing subsequent health risk for young victims of intentional injuries and their families, the violence reduction effort will address the following objectives:

* Develop detailed profiles of participants treated at the Pediatric Emergency Department through a detailed behavior and attitude assessment battery given in an interview format. Additionally, this information will be used to increase understanding of the needs of this at-risk population for the purpose of developing preventive services. Data from these assessments will also be used in the preparation of scholarly papers on this patient population and the impact of this program on their recidivism.
* Provide brief violence prevention (BVP) intervention to youth to review conflict-resolution strategies, increase their awareness of youth's risk factors for recidivism, explore coping skills, and develop safety plan services and supports that may be responsive to their needs and reduce the likelihood of future risk of intentional injury.
* Provide brief violence awareness (BVA) intervention to provide basic information on the prevalence, impact of violence and the available community resources.
* Provide comprehensive case management to participants in order to maintain program involvement.
* Provide a curriculum consisting of skill building, educational development, increased exposure to health careers and internship opportunities.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Reside in the 23223 zip code of the City of Richmond
2. Attend Martin Luther King Middle School
3. Be between the ages 10-15.

Exclusion Criteria:

* Not being fluent in English
* Developmental and cognitive delays or any other type of physical or mental problems that would prevent them from answering interview questions or participating
* Experiencing child abuse
* Being identified or documented as experiencing suicidal or homicidal ideation, predatory sexual behavior or perpetration of violent behavior
* Violent behavior towards staff and/or other patients

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
Behaviors and attitudes related to violence - assessment consisting of select questions from various tools. | Every nine weeks up to seven years, from study enrollment through graduation from high school or participants' voluntary withdrawal from the study, whichever comes first.
  The assessment contains select questions from the following: Future Aspirations - Peer Leader Survey, Rochester Youth Development Study, Individual Protective Factor Index, Center for Epidemiological Studies Depression Scale for Children, Attitude Toward Interpersonal Peer Violence Scale, Children's Exposure to Community Violence Scale, Self-Reported Delinquency Problem Behavior Frequency Scale, and CDC Youth Risk Behavior Surveillance System.

SECONDARY OUTCOMES:
Reduction in the number of violence related hospital visits | Annually for the duration of this study, up to seven years.
Reduction in violence related activities that led to hospital visits or delinquent behavioral involvement | Annually for the duration of this study, up to seven years.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Aboutanos, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - MLK Middle School Boys and Girls Club, Richmond, Virginia
  - VCU Pediatric Emergency Department, Richmond, Virginia